CLINICAL TRIAL: NCT03739281
Title: Advancing Diagnosis and Treatment for Lung Cancer Patients Using Hybrid PET/MR Imaging and Novel Visualization Tools
Brief Title: PET/MR Imaging in Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Internal resources ended
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/1952
Record Dates: First submitted 2018-10-30; First posted 2018-11-13 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nuclear medicine imaging (Other): Patients undergo nuclear medicine imaging with PET/MR and PET/CT.
  Interventions: Diagnostic Test: PET/MR; Diagnostic Test: PET/CT

INTERVENTIONS:
Diagnostic Test: PET/MR — The included patients are imaged with PET/MR as part of the research protocol.
Diagnostic Test: PET/CT — The included patients are imaged with PET/CT as part of normal clinical routine.

SUMMARY:
The purpose of this project is to investigate if PET/MR imaging improves the accuracy in visualization and characterization of lung cancer disease, compared to PET/CT.

DETAILED DESCRIPTION:
Lung cancer is the most frequent cancer type and the leading cause of cancer-related death worldwide. Positron emission tomography (PET) coupled with computed tomography (CT) is the standard of care for visualization and staging of lung cancer. Recent clinical introduction of hybrid PET and magnetic resonance (MR) imaging systems has shown potential to improve tumor imaging beyond the limits of PET/CT. However, knowledge about the clinical impact of this new hybrid modality is still limited.

This project aims to investigate how PET/MR may improve the diagnosis and treatment of lung cancer disease, compared to PET/CT: PET/MR may allow early detection of brain and liver metastases, which strongly affects treatment outcome and survival; predictive models based on machine learning may combine image derived biomarkers from PET/MR, histology and health record data, to automatically visualize and characterize the tumor, facilitating computer aided diagnosis and personalized radiotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Referred to clinical PET/CT examination for investigation of lung disease.

Exclusion Criteria:

* Blood glucose level >8.3 mmol/l
* MR incompatible objects, e.g. metal implants, inside the body
* Intolerance to gadolinium-based contrast agents, e.g. severe renal disease (GFR<30).
* Unable to give written consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of PET/MR vs. clinical routine PET/CT | 1-2 weeks after the initial inclusion.
  Sensitivity and specificity of PET/MR scans will be compared with in clinical routine PET/CT examinations for lung cancer disease feature prediction.

SECONDARY OUTCOMES:
Prediction of treatment response and progression-free survival | 1 year after inclusion.
  We will investigate which PET/MR or PET/CT features are best suited as an imaging biomarker for treatment response evaluation and for progression-free survival 1 year after inclusion.
Prediction of treatment response and progression-free survival | 2 years after inclusion.
  We will investigate which PET/MR or PET/CT features are best suited as an imaging biomarker for treatment response evaluation and for progression-free survival 2 years after inclusion.
Prediction of treatment response and progression-free survival | 5 years after inclusion.
  We will investigate which PET/MR or PET/CT features are best suited as an imaging biomarker for treatment response evaluation and for progression-free survival 5 years after inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Rune Sundset, MD, PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway